CLINICAL TRIAL: NCT05901155
Title: Impact of medAL-mentor, a Real-time Mentoring and Benchmarking Tool, on Antibiotic Prescription Among Children in Primary Health Care Facilities in Tanzania
Brief Title: Impact of a Real-time Mentoring Tool on Antibiotic Prescription (medAL-mentor)
Acronym: medAL-mentor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Ifakara Health Institute (Other); Mbeya Medical Research Centre-National Institute for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-02800_substudymedalmentor
Record Dates: First submitted 2023-05-11; First posted 2023-06-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Primary Health Care for Children
Keywords: Digital health; Antibiotic stewardship; Real-time mentoring; Benchmarking; Clinical decision support algorithm

STUDY DESIGN:
Intervention Model Description: The study involves two arms: intervention and control. Health facilities will serve as clusters, with half of the facilities (20) receiving the intervention and the other half serving as controls (20). Health facilities will be randomized to their respective study arm. A parallel design (all health facilities start at the same time) will be used.
Masking Description: Masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MedAL-mentor (Experimental): In health facilities allocated to the medAL-mentor arm, the intervention will consist in :
  * Providing tablets with ePOCT+ and initial training for use by healthcare workers
  * Access to medAL-mentor for healthcare workers and the monitoring team
  * Regular (at least every 2 weeks) supportive messages sent by the monitoring team to healthcare workers providing feedback from medAL-mentor
  * Targeted phone calls and health facilities visits by the monitoring team based on medAL-mentor review Monitoring will be performed by the study team.
  Interventions: Device: MedAL-mentor
- Routine mentoring (No Intervention): In health facilities allocated to the control arm, tablets with ePOCT+ will also be provided to healthcare workers with initial training, but subsequent mentoring will be conducted routinely:
  * No access to medAL-mentor for healthcare workers or the monitoring team
  * At least one message sent by the monitoring team to healthcare workers every two weeks, to inquire about any issues and trigger a site visit if needed
  * At least one visit from the monitoring team in each health facility every two months Monitoring will be performed by the study team.

INTERVENTIONS:
Device: MedAL-mentor — MedAL-mentor is a near real-time monitoring and benchmarking dashboard based on data collected through ePOCT+, providing direct feedback on several clinical indicators (antibiotic prescription, performance of key measurements, signs, and diagnostic tests).
  Arms: MedAL-mentor

SUMMARY:
The goal of this ancillary study, part of the DYNAMIC project, is to reduce antibiotic prescription and improve the quality of care for children in primary care in Tanzania using a near real-time mentoring tool (called medAL-mentor), based on a monitoring and benchmarking dashboard and feedback by the monitoring team. The main question to be answered is: Can real-time mentoring, based on clinical decision support algorithm data, improve healthcare workers' compliance with guidelines - and therefore quality of care for paediatric outpatients? Health providers in participating health facilities will receive either the medAL-mentor tool and feedback from the monitoring team (intervention group), or standard mentoring (control group), so that the impact on antibiotic prescription and other quality of care indicators can be compared between the two arms.

DETAILED DESCRIPTION:
ePOCT+ is a paediatric digital clinical decision support algorithm for health workers in primary care facilities in Tanzania. The objective is to improve the integrated management of acutely ill children aged 1 day to 14 years and reduce inappropriate antibiotic prescriptions.

Preliminary findings from the first phase of the DYNAMIC project, an open-label cluster randomized controlled study performed in 40 health facilities, showed a reduction in antibiotic prescription by health providers from about 70% in the control arm to 23% in health facilities using ePOCT+, with similar clinical outcomes in children at day 7. Nevertheless, uptake of ePOCT+ and antibiotic prescription in the intervention arm were very heterogeneous across health facilities.

Benchmarking in healthcare is defined as "a process of comparative evaluation and identification of the underlying causes leading to high levels of performance". The findings and experiences of different institutions are shared, and elements of best practices are adopted to improve performance. Benchmarking has been promoted for years by infectious diseases societies as a component of hospital antimicrobial stewardship programs, to reduce antibiotic prescription. Benchmarking has also been shown to be an effective incentive to improve the quality of care in various settings, including primary care practice. Unfortunately, published initiatives have largely come from high-income countries.

In the context of the DYNAMIC project, we developed a near real-time mentoring tool, medAL-mentor, based on a monitoring and benchmarking dashboard using data collected through ePOCT+. The tool provides direct feedback to health workers on their performance, based on several clinical indicators (including antibiotic prescription), in comparison with data from other health facilities. The monitoring team will target calls and monitoring visits to health facilities based on these indicators and use the dashboard to facilitate discussions with healthcare workers.

This ancillary study, MedAL-mentor, aims to assess whether this real-time mentoring tool based on data generated by a clinical decision support algorithm, as well as feedback from the mentoring team, improves healthcare workers' compliance with guidelines - and therefore the quality of care for sick children at primary care level.

More specifically, the study objectives are :

Primary objective :

To determine whether the provision of medAL-mentor, a digital mentoring tool, decreases antibiotic prescription by primary care clinicians using a clinical decision support algorithm (ePOCT+) for the management of sick children

Secondary objectives are :

1. To assess the impact of medAL-mentor on clinicians' uptake of ePOCT+
2. To assess the impact of medal-mentor on clinicians in terms of :

   1. Performance of key measurements and assessment of signs by clinicians
   2. Compliance with the recommendations related to point-of-care tests (for malaria and haemoglobin)

This open-label, parallel cluster randomized controlled study is embedded in the second phase of the DYNAMIC project in Tanzania. The intervention consists of providing direct access to medAL-mentor to the healthcare workers. The mentoring team will target calls and monitoring visits to health facilities based on medAL-mentor indicators and use the dashboard to facilitate discussions with healthcare workers during the monitoring visits. Since the intervention takes place at the healthcare worker level and their practices are influenced by the context of the health facility they are working in, randomization at the health facility level rather than at the health worker level was chosen.

40 health facilities using ePOCT+ for the first time during the second phase of the DYNAMIC project will be randomly selected and assigned to two groups (randomization 1:1, intervention: control). Health workers in health facilities randomized to the intervention group will receive feedback on their performance through direct access to medAL-mentor and regular mobile messages, as well as targeted phone calls and visits by the monitoring team based on the medAL-mentor dashboard. Health facilities from the control group will receive standard monitoring (regular messages to check for any issues and regular site visits), without access to medAL-mentor (neither for the health workers nor for the monitoring team).

ELIGIBILITY:
Inclusion Criteria:

- Presenting for an acute medical or surgical condition

Exclusion Criteria:

* Presenting for scheduled consultation for a chronic disease (e.g. HIV, tuberculosis, non-communicable diseases, malnutrition)
* Presenting for routine preventive care (e.g. growth monitoring, vitamin supplementation, deworming, vaccination)

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37000 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of children prescribed an antibiotic in the intervention group (medAL-mentor) as compared to the control group (routine mentoring) | Day 0 (by the end of the consultation)
  Number of children for whom at least one systemic (oral or parenteral) antibiotic has been prescribed during consultation, over all eligible children, as reported by the healthcare workers in a routine registry

SECONDARY OUTCOMES:
Percentage of consultations with eligible children performed using ePOCT+ | Day 0 (by the end of the consultation)
  Number of consultations completed with ePOCT+, over all consultations with eligible children as reported in a routine registry
Percentage of children in whom key signs have been checked by healthcare workers | Day 0 (by the end of the consultation)
  Number of children in whom key signs (temperature, weight, mid-upper arm circumference (MUAC), respiratory rate) have been checked by healthcare workers, over the total number of children for whom this was recommended, as reported by healthcare workers in ePOCT+
Percentage of children for whom appropriate diagnostic tests have been performed by healthcare workers | Day 0 (by the end of the consultation)
  Number of children for whom diagnostic tests (haemoglobin and malaria tests) have been performed by healthcare workers, over the total number of children for whom diagnostic tests were recommended, as reported by healthcare workers in ePOCT+

CONTACTS AND LOCATIONS:
Locations (40):
- Tanzania (40):
  - Idiga Dispensary, Idiga, Mbeya
  - Igoma Dispensary, Igoma, Mbeya
  - Lwanjilo Dispensary, Ilowelo, Mbeya
  - Inyala Health Center, Inyala, Mbeya
  - Iwindi Dispensary, Iwindi, Mbeya
  - Kimondo Dispensary, Kimondo, Mbeya
  - Mbalizi Dispensary, Mbalizi, Mbeya
  - Mjele Dispensary, Mjele, Mbeya
  - Mshewe Dispensary, Mjele, Mbeya
  - Mwabwowo Dispensary, Mwabwowo, Mbeya
  - Santilya Health Center, Santilya, Mbeya
  - Shuwa Dispensary, Shuwa, Mbeya
  - Songwe viwandani Dispensary, Songwe, Mbeya
  - Chikuti Dispensary, Chikuti, Morogoro
  - Chirombora Dispensary, Chirombora, Morogoro
  - Chita Rural Dispensary, Chita, Morogoro
  - Idete Dispensary, Idete, Morogoro
  - Idunda Dispensary, Idunda, Morogoro
  - Kibaoni Health Center, Ifakara, Morogoro
  - Michenga Dispensary, Ifakara, Morogoro
  - Sagamaganga Dispensary, Ifakara, Morogoro
  - Ketaketa Dispensary, Kataketa, Morogoro
  - Kichangani Dispensary, Kichangani, Morogoro
  - Kisegese Dispensary, Kisegese, Morogoro
  - Mbuga Dispensary, Mbuga, Morogoro
  - Milola Dispensary, Milola, Morogoro
  - Mngeta Health Center, Mngeta, Morogoro
  - Sanje Dispensary, Sonjo, Morogoro
  - Sonjo Dispensary, Sonjo, Morogoro
  - Udagaji Dispensary, Udagaji, Morogoro
  - Utengule Dispensary, Utengule, Morogoro
  - Isyesye Dispensary, Mbeya
  - Itagano Dispensary, Mbeya
  - Itensa Dispensary, Mbeya
  - Itezi Dispensary, Mbeya
  - Itijy Dispensary, Mbeya
  - Iyunga Health Center, Mbeya
  - Ndanyela Dispensary, Mbeya
  - Nzovwe Health Center, Mbeya
  - Tembela Dispensary, Mbeya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis J. All inclusive benchmarking. J Nurs Manag. 2006 Jul;14(5):377-83. doi: 10.1111/j.1365-2934.2006.00596.x. PMID 16787472
- [Background] Thonon F, Watson J, Saghatchian M. Benchmarking facilities providing care: An international overview of initiatives. SAGE Open Med. 2015 Sep 23;3:2050312115601692. doi: 10.1177/2050312115601692. eCollection 2015. PMID 26770800
- [Background] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Background] Willmington C, Belardi P, Murante AM, Vainieri M. The contribution of benchmarking to quality improvement in healthcare. A systematic literature review. BMC Health Serv Res. 2022 Feb 2;22(1):139. doi: 10.1186/s12913-022-07467-8. PMID 35109824
- [Background] Piccoliori G, Mahlknecht A, Abuzahra ME, Engl A, Breitenberger V, Vogele A, Montalbano C, Sonnichsen A. Quality improvement in chronic care by self-audit, benchmarking and networking in general practices in South Tyrol, Italy: results from an interventional study. Fam Pract. 2021 Jun 17;38(3):253-258. doi: 10.1093/fampra/cmaa123. PMID 33184661
- [Background] Hermans MP, Elisaf M, Michel G, Muls E, Nobels F, Vandenberghe H, Brotons C; OPTIMISE International Steering Committee. Benchmarking is associated with improved quality of care in type 2 diabetes: the OPTIMISE randomized, controlled trial. Diabetes Care. 2013 Nov;36(11):3388-95. doi: 10.2337/dc12-1853. Epub 2013 Jul 11. PMID 23846810
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- See also: Dynamic study website — https://dynamic-study.com/

DOCUMENTS (2):
  • Study Protocol (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT05901155/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT05901155/SAP_001.pdf